CLINICAL TRIAL: NCT03080064
Title: Supporting Healthful Lifestyles During Pregnancy: A Health Coach Intervention Pilot Study
Brief Title: Health Coach Intervention Pilot Study
Acronym: AHA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard Pilgrim Health Care (Other)
Collaborators: American Heart Association (Other); Harvard Vanguard Medical Associates (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PH000523C; 14CRP20490354 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2017-02-22; First posted 2017-03-15 (Actual); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: Satisfaction
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: One-arm intervention trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health Coach Intervention (Experimental): The investigators connected participants at enrollment (median gestation of 12.5 weeks, IQR: 11-15) with a trained health coach who called participants every 2-3 weeks until 36 weeks of gestation. During these phone calls, health coaches helped participants adopt and maintain new healthful lifestyle behaviors that were evidence-based, simple, and easy to track. Goals aimed to promote appropriate gestational weight gain and covered several domains including diet, physical activity, screen time, and sleep.
  Interventions: Behavioral: Health Coach Intervention

INTERVENTIONS:
Behavioral: Health Coach Intervention — Please see arm description.

SUMMARY:
In this mixed methods study, the investigators assessed the feasibility and acceptability of a remote health coach intervention to promote healthful lifestyle behaviors among overweight pregnant women. At one northeastern US clinic, the investigators enrolled 30 overweight (pre-pregnancy BMI≥25 kg/m2) pregnant women at a median gestation of 12.5 weeks (IQR: 11-15) into a one arm intervention trial. The investigators connected participants with a health coach to provide behavioral support to help participants adopt or maintain healthy lifestyle goals during pregnancy. Health coaches contacted participants by phone every 2-3 weeks to monitor goals, and sent emails and text messages to check-in between calls. To assess the intervention, participants completed baseline (N=30) and follow-up surveys at the end of the intervention (N=26), as well as follow-up phone interviews (N=18).

DETAILED DESCRIPTION:
<Health Coach Intervention > The investigators connected participants at enrollment (median gestation of 12.5 weeks, IQR: 11-15) with a trained health coach who called participants every 2-3 weeks until 36 weeks of gestation. During these phone calls, health coaches helped participants adopt and maintain new healthful lifestyle behaviors that were evidence-based, simple, and easy to track. Goals aimed to promote appropriate gestational weight gain and covered several domains including diet, physical activity, screen time, and sleep.

During the first call, health coaches invited participants to prioritize these goals according to their level of self-efficacy, readiness to change, preferences, and values. Throughout the intervention, health coaches used principles of motivational interviewing that relied on a patient-centered approach to enhance readiness to change by exploring ambivalence and resistance to change. In addition to setting personal goals, health coaches also presented optimal goals for ideal cardiovascular health.

During follow-up calls, health coaches monitored progress and helped adjust goals when necessary (e.g. too many goals, or the goal was too ambitious). Health coaches also addressed barriers and potential solutions with participants, and helped them target higher goal settings or select novel goals when participants attained them. Health coaches sent emails or text messages depending on participant preferences to check-in about progress toward goals or clinical appointments between calls. Research staff (including an MD) met weekly with health coaches to review their conversations with participants, and to address any medical issues to ensure that it would be reported to the primary care provider obstetric team if appropriate.

<Study Design and Sample> Participants completed baseline (N=30) and follow-up (N=26) surveys at the end of the intervention as well as follow-up phone interviews (N=18). Surveys collected information on demographics, attitudes related to weight status and pregnancy, opinions about the intervention, and included food frequency questions . Interviews followed a guide of open-ended questions to determine insights on what helped achieve goals, motivation, opinions of the health coach intervention, and areas for improvement. One study staff member, who has experience with qualitative data collection, conducted all of the individual interviews. This study was approved by the Harvard Pilgrim Health Care Human Studies Committee.

ELIGIBILITY:
Inclusion Criteria:

* pregnant (less than 16 weeks of gestation),
* overweight or obese (pre-pregnancy BMI≥25 kg/m2),
* 18 years of age or older,
* English speaking,
* planned to remain at the same obstetrics clinic for the duration of their pregnancies.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-07-16 (Actual); Primary Completion 2016-06-27 (Actual); Study Completion 2016-06-27 (Actual)

PRIMARY OUTCOMES:
Satisfaction with the health coach intervention as assessed by surveys | From enrollment until the end of the intervention at 36 weeks of gestation.
  The investigators assessed the feasibility and acceptability of a remote health coach intervention to promote healthful lifestyle behaviors among overweight pregnant women using baseline and follow-up surveys.
Satisfaction with the health coach intervention as assessed by phone interviews | From enrollment until the end of the intervention at 36 weeks of gestation.
  Using an interview guide, the investigators assessed the feasibility and acceptability of a remote health coach intervention to promote healthful lifestyle behaviors among overweight pregnant women.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-France Hivert, MD, MMSc, Principal Investigator — Harvard Pilgrim Health Care Institute
Locations (1):
- Harvard Pilgrim Health Care Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Seward MW, Simon D, Richardson M, Oken E, Gillman MW, Hivert MF. Supporting healthful lifestyles during pregnancy: a health coach intervention pilot study. BMC Pregnancy Childbirth. 2018 Sep 17;18(1):375. doi: 10.1186/s12884-018-2010-z. PMID 30223779